CLINICAL TRIAL: NCT00393796
Title: Randomized Blinded Phase II Trial of Maintenance SUO11248 Versus Placebo Post Chemotherapy for Patients With Advanced Urothelial Carcinoma
Brief Title: Trial of Maintenance SUO11248 Versus Placebo Post Chemotherapy for Patients With Advanced Urothelial Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UMCC 2005.145; NCT01225848 (obsolete NCT alias)
Record Dates: First submitted 2006-10-27; First posted 2006-10-30 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SUTENT (Active Comparator): Study participants randomized to received SUTENT will receive a dose of 50 mg PO (capsules) as a single agent to be taken once daily for four consecutive weeks followed by a two week rest period to form a complete cycle of six weeks.
  Interventions: Drug: SUTENT
- Placebo (Placebo Comparator): Study participants randomized to receive placebo will receive 50 mg/day PO (capsules) of an inactive substance to be taken once daily for four consecutive weeks followed by a two week rest period to form a complete cycle of six weeks.
  Interventions: Drug: SUTENT; Other: Placebo

INTERVENTIONS:
Drug: SUTENT — 50 mg/PO once daily for four consecutive weeks with a two week rest period. Study participants who show evidence of disease progression (or are considered for removal from study for any other reason) will be unblinded. Participants receiving SU011248 will be removed from the study. Participants receiving placebo will be given the opportunity to "crossover" and receive SU011248.
  Other Names: SU011248
Other: Placebo
  Arms: Placebo

SUMMARY:
This study is a randomized, blinded, placebo-controlled study evaluating the drug, SUO11248 (SUTENT), for maintenance therapy in advanced urothelial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologic/cytologic diagnosis of urothelial carcinoma (transitional cell carcinoma either pure or mixed histology)
* All patients must have received four - six cycles of standard first line chemotherapy (protocol details suggested combinations) for treatment of locally recurrent or metastatic disease AND must have achieved stable disease (SD), partial response (PR), or complete response (CR) to this chemotherapy.
* Type of response, number of cycles and specific regimen given must be carefully recorded and submitted at time of registration.
* Reports from pre and post treatment imaging will be required at time of registration to document response.
* Patients must be registered within 1 month (or the next business day if falls on a weekend or holiday) of scans demonstrating stable disease or better and no more than 42 days after receiving the last standard chemotherapy dose. For example, if patients are receiving treatment on days 1 and 8 of each cycle, day 8 of the last cycle would be considered the last standard chemotherapy dose.
* Patients may have received previous adjuvant or neoadjuvant therapy.
* No prior antiangiogenic therapy for this stage of the disease.

Exclusion Criteria:

* Major surgery within 4 weeks of starting the study treatment.
* NCI CTCAE grade 3 hemorrhage or higher within 4 weeks of starting the study treatment.
* History of or known spinal cord compression, or carcinomatous meningitis, or evidence of symptomatic brain or leptomeningeal disease on screening CT or MRI scan. However treated, stable and asymptomatic brain metastases are allowed.
* Known HIV - positive patients may not participate. This is to avoid additional complications that immune suppression and HIV infection may cause due to the intense nature of the chemotherapy in this trial.
* Any of the following within 6 months prior to study administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (CHF), cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Patients with history of or who are suspected to have CHF can be included as long as they are asymptomatic and have an ejection fraction that is equal to or above the institutional lower limit of normal by baseline MUGA(obtained within one month of registration or the next business day if falls on a weekend or holiday).
* Ongoing cardiac dysrhythmias of NCI CTCAE Grade > 2.
* Unresolved bacterial infection.
* Uncontrolled hypertension.
* Pre-existing thyroid abnormality that can not be controlled medically.
* Concurrent treatment on another clinical trial.
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-05; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maha H. Hussain, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (9):
- United States (9):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - The University of Chicago, Chicago, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Weill Medical College of Cornell University, New York, New York
  - Columbia University Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Result] Grivas PD, Daignault S, Tagawa ST, Nanus DM, Stadler WM, Dreicer R, Kohli M, Petrylak DP, Vaughn DJ, Bylow KA, Wong SG, Sottnik JL, Keller ET, Al-Hawary M, Smith DC, Hussain M. Double-blind, randomized, phase 2 trial of maintenance sunitinib versus placebo after response to chemotherapy in patients with advanced urothelial carcinoma. Cancer. 2014 Mar 1;120(5):692-701. doi: 10.1002/cncr.28477. Epub 2013 Nov 18. PMID 24249435

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were originally randomized to SUTENT or Placebo (Double Blind Period). 26 participants were randomized to SUTENT. Of the 28 participants randomized to Placebo, those that progressed were offered SUTENT if they were eligible.
Period: Double Blind Period
Arm/Group | SUTENT | Placebo
Started | 26 | 28
Completed | 26 | 28
Not Completed | 0 | 0
Period: Open Label Period - Placebo to SUTENT
Arm/Group | SUTENT | Placebo
Started | 0 | 16
Completed | 0 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SUTENT | Placebo | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Continuous [Median (Full Range); unit: years] | 69 [48 to 84] | 69 [53 to 81] | 69 [48 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 20 | 19 | 39
ECOG Performance Status [Number; unit: participants] — The Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) is a measure of general well being and activities of daily life. Scores run from 0 to 5 where 0 denotes normal activity and 5 represents death.
  participants
    PS=0 | 10 | 11 | 21
    PS=1 | 15 | 17 | 32
    PS=2 | 1 | 0 | 1
Visceral Metastasis [Number; unit: participants] — The number of participants presenting with visceral metastasis.
  participants | 9 | 12 | 21
Bladder Primary Tumor [Number; unit: participants] — The number of participants presenting with primary bladder tumors.
  participants | 20 | 18 | 38
Mixed Histology [Number; unit: participants] — The number of participants presenting with mixed histology.
  participants | 2 | 4 | 6
Prior Chemotherapy Regimen [Number; unit: participants] — The number of participants that had the following prior chemotherapy regimens: Cisplatin and gemcitabine, MVAC (methotrexate, vinblastine, doxorubicin and cisplatin), Non-cisplatin-containing chemotherapy.
  participants
    Cisplatin and gemcitabine | 10 | 14 | 24
    MVAC | 3 | 2 | 5
    Non-cisplatin-containing chemotherapy | 13 | 12 | 25
Response to Prior Chemotherapy [Number; unit: participants] — The number of participants that experienced the following best overall response from prior chemotherapy: CR (Complete Response), PR (Partial Response), and SD (Stable Disease).
  participants
    CR | 3 | 1 | 4
    PR | 10 | 12 | 22
    SD | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Experience Progression by 6 Months for Participants Receiving Sunitinib and Participants Receiving Placebo
Description: The primary endpoint of this unblinded, randomized trial is to compare the 6-month progression rate in patients randomized to maintenance SU011248 as compared with placebo following primary chemotherapy.
  Progression is defined as a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 6 Months Post Treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SUTENT | Placebo
Number analyzed (Participants) | 26 | 28
percentage of participants | 71.7 [54 to 87] | 64.3 [47 to 81]

ADVERSE EVENTS:
Groups:
- SUTENT: Study participants randomized to received SUTENT will receive a dose of 50 mg PO (capsules) as a single agent to be taken once daily for four consecutive weeks followed by a two week rest period to form a complete cycle of six weeks.
  26 participants were randomized to SUTENT and 16 participants randomized to Placebo crossed over to SUTENT during treatment so a total of 42 participants were treated with SUTENT.
- Placebo Only: Study participants randomized to receive placebo will receive 50 mg/day PO (capsules) of an inactive substance to be taken once daily for four consecutive weeks followed by a two week rest period to form a complete cycle of six weeks.
  28 participants were randomized to Placebo. 16 of these 28 patients later received SUTENT.
Arm/Group | SUTENT | Placebo Only
Serious Adverse Events (participants affected / at risk) | 17/42 | 6/28
Other Adverse Events (participants affected / at risk) | 42/42 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SUTENT (N=42) | Placebo Only (N=28)
Cardiac General - Other (Cardiac disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Death not associated with CTCAE term (General disorders) | 5 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 | 1
Hemoglobin (Blood and lymphatic system disorders) | 2 | 1
Hemorrhage, GI (Vascular disorders) | 1 | 1
Infection with Grade 3 or 4 neutrophils (Infections and infestations) | 2 | 1
Infection with unknown ANC (Infections and infestations) | 1 | 1
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Obstruction, GI (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 1 | 2
Platelets (Blood and lymphatic system disorders) | 2 | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 | 0
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Syncope (fainting) (Nervous system disorders) | 1 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 1
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 | 1
CNS cerebrovascular ischemia (Vascular disorders) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 0 | 1
Obstruction, GU (Renal and urinary disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SUTENT (N=42) | Placebo Only (N=28)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 6 | 4
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 11 | 5
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5 | 3
Alkaline phosphatase (Investigations) | 4 | 5
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 20 | 12
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 3 | 1
Ataxia (incoordination) (Nervous system disorders) | 1 | 1
Blood/Bone Marrow - Other (Specify) (Blood and lymphatic system disorders) | 1 | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 | 1
CD4 count (Investigations) | 3 | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 6 | 4
Cardiac Arrhythmia - Other (Specify) (Cardiac disorders) | 1 | 1
Cardiac General - Other (Specify) (Cardiac disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Confusion (Nervous system disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 15 | 11
Constitutional Symptoms - Other (General disorders) | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Creatinine (Investigations) | 15 | 11
Cystitis (Renal and urinary disorders) | 5 | 3
Death not associated with CTCAE term (General disorders) | 5 | 3
Dehydration (Metabolism and nutrition disorders) | 7 | 3
Dermatology/Skin - Other (Specify) (Skin and subcutaneous tissue disorders) | 9 | 2
Diarrhea (Gastrointestinal disorders) | 24 | 12
Distension/bloating, abdominal (Gastrointestinal disorders) | 5 | 3
Dizziness (Nervous system disorders) | 7 | 11
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 4 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 2
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Edema: head and neck (General disorders) | 4 | 2
Edema: limb (General disorders) | 5 | 6
Endocrine - Other (Endocrine disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 30 | 23
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <'1.0 x 10e9/L) (General disorders) | 5 | 3
Flatulence (Gastrointestinal disorders) | 4 | 1
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 4 | 1
Gastrointestinal - Other (Gastrointestinal disorders) | 1 | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 10 | 11
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 | 1
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 6 | 5
Hearing: patients with/without baseline audiogram and enrolled in a monitoring program (Ear and labyrinth disorders) | 1 | 1
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 2 | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 | 3
Hematoma (Vascular disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 18 | 13
Hemoglobinuria (Blood and lymphatic system disorders) | 1 | 0
Hemorrhage, GI (Vascular disorders) | 3 | 2
Hemorrhage, GU (Vascular disorders) | 9 | 5
Hemorrhage, pulmonary/upper respiratory (Vascular disorders) | 5 | 1
Hemorrhage/Bleeding - Other (Specify) (Vascular disorders) | 3 | 2
Hemorrhoids (Gastrointestinal disorders) | 3 | 1
Hot flashes/flushes (Vascular disorders) | 1 | 0
Hyperbilirubinemia (Investigations) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Cardiac disorders) | 14 | 10
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 1
Hypotension (Cardiac disorders) | 2 | 1
Incontinence, anal (Gastrointestinal disorders) | 1 | 0
Incontinence, urinary (Renal and urinary disorders) | 2 | 2
Infection with Grade 3 or 4 neutrophils (Infections and infestations) | 4 | 4
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 5 | 3
Infection with unknown ANC (Infections and infestations) | 3 | 3
Injection site reaction/extravasation changes (General disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 3 | 2
Joint-function (Musculoskeletal and connective tissue disorders) | 1 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 2
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 13 | 6
Leukopenia (Blood and lymphatic system disorders) | 4 | 2
Lipase (Metabolism and nutrition disorders) | 1 | 0
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 | 0
Lymphatics - Other (Vascular disorders) | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 6 | 3
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 2 | 1
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 4 | 1
Memory impairment (Nervous system disorders) | 3 | 3
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 3 | 2
Mood alteration (Psychiatric disorders) | 2 | 1
Mucositis/stomatitis (clinical exam) (Investigations) | 5 | 0
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 6 | 1
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 8 | 5
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 17 | 11
Neurology - Other (Nervous system disorders) | 2 | 2
Neuropathy: cranial (Nervous system disorders) | 1 | 0
Neuropathy: motor (Nervous system disorders) | 4 | 2
Neuropathy: sensory (Nervous system disorders) | 13 | 6
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 6 | 7
Obstruction, GI (Gastrointestinal disorders) | 1 | 1
Obstruction/stenosis of airway (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PTT (Partial Thromboplastin Time) (Investigations) | 2 | 0
Pain (General disorders) | 42 | 28
Pain - Other (General disorders) | 9 | 8
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 | 0
Platelets (Blood and lymphatic system disorders) | 24 | 10
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 4 | 2
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 2 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4 | 2
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 1 | 1
Pulmonary/Upper Respiratory - Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 10 | 6
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 7 | 3
Renal failure (Renal and urinary disorders) | 2 | 1
Renal/Genitourinary - Other (Renal and urinary disorders) | 3 | 2
Rigors/chills (General disorders) | 6 | 4
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 7 | 3
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2 | 0
Sweating (diaphoresis) (General disorders) | 2 | 1
Syncope (fainting) (Nervous system disorders) | 3 | 2
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 13 | 6
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 2
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 1 | 0
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 6 | 5
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Tremor (Nervous system disorders) | 2 | 1
Ulceration (Skin and subcutaneous tissue disorders) | 3 | 1
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 4 | 8
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 | 1
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 | 1
Vision-blurred vision (Eye disorders) | 1 | 0
Vitreous hemorrhage (Vascular disorders) | 1 | 0
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 11 | 6
Watery eye (epiphora, tearing) (Eye disorders) | 2 | 0
Weight loss (General disorders) | 5 | 2
CNS cerebrovascular ischemia (Vascular disorders) | 0 | 1
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 | 1
Dermal change lymphedema, phlebolymphedema (Skin and subcutaneous tissue disorders) | 0 | 1
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 0 | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
INR (International Normalized Ratio of prothrombin time) (Investigations) | 0 | 1
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 | 1
Obstruction, GU (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Infections and infestations) | 0 | 1
Vaginal dryness (Reproductive system and breast disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This multicenter study was limited by premature closure and a small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes